CLINICAL TRIAL: NCT02561429
Title: Comparison of Difference Histamine Concentration (1, 5 and 10 mg/ml) for Positive Control of Skin Prick Test
Brief Title: Comparison of Difference Histamine Concentration (1, 5 and 10 mg/ml) for Skin Prick Test Positive Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Prof, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: si645/2012
Record Dates: First submitted 2015-09-15; First posted 2015-09-28 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Immediate Hypersensitivity
MeSH Terms: conditions — Hypersensitivity, Immediate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SPT of histamine (Experimental): SPT of histamine concentration 1, 5 and 10 mg/ml
  Interventions: Procedure: SPT

INTERVENTIONS:
Procedure: SPT — SPT of histamine concentration 1, 5 and 10 mg/ml

SUMMARY:
Skin prick test (SPT) was used for diagnostic test for type 1 hypersensitivity. The efficacy and safety of SPT were proved. The positive control of SPT is histamine.

In Thailand, the most common concentration of histamine for SPT is 10 mg/ml. However, in some practice they use other concentration (1, 2.5 mg/ml).

This study will find the proper concentration of histamine for positive control use in SPT.

DETAILED DESCRIPTION:
Appropriate concentration of histamine positive control is important in interpretation the result of skin prick test.

ELIGIBILITY:
Inclusion Criteria:

* Parcitipate person who attented allergy clinic, ENT clinic
* Legible in Thai language

Exclusion Criteria:

* Patient cannot withhold antihistamine drug
* Pragnancy and lactation mother
* comorbid disease such as cardiac disease, liver, renal, hypertension and severe asthma

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Mean wheal diameters of SPT of different histamine concentrations. | 1 years
  compare mean wheal diameters of histamine concentration 1,5, and 10 mg/ml

SECONDARY OUTCOMES:
Mean wheal diameters of SPT of local and imported histamine positive concentration | 1 year
  compare mean wheal diameters of imported histamine 1 mg/ml to local histamine

CONTACTS AND LOCATIONS:
Overall Officials: Nualanong Visitsunthorn, Prof, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Menardo JL, Bousquet J, Rodiere M, Astruc J, Michel FB. Skin test reactivity in infancy. J Allergy Clin Immunol. 1985 Jun;75(6):646-51. doi: 10.1016/0091-6749(85)90088-0. PMID 2409121
- [Result] Berkowitz RB, Tinkelman DG, Lutz C, Crummie A, Smith K. Evaluation of the Multi-Test device for immediate hypersensitivity skin testing. J Allergy Clin Immunol. 1992 Dec;90(6 Pt 1):979-85. doi: 10.1016/0091-6749(92)90471-d. PMID 1460201